CLINICAL TRIAL: NCT06807554
Title: Intraperitoneal Ketamine Versus Bupivacaine for Postoperative Pain Control After Laparoscopic Cholecystectomy
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Liaquat National Hospital & Medical College (Other)
Responsible Party: Principal Investigator, Shehrum Bughio, Principal investigator, Liaquat National Hospital & Medical College
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Liaquat National Hospital
Record Dates: First submitted 2025-01-29; First posted 2025-02-04 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Laparoscopic Cholecystectomy Surgery
Keywords: Laparoscopic surgery; Ketamine; Bupivacaine; Intraperitoneal instillation; Cholecystectomy
MeSH Terms: interventions — Ketamine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group K (Experimental): In Group K, ketamine 0.25mg/kg diluted in normal saline to a total volume of 40 ml was instilled by the surgeon, 20 ml before starting gall bladder dissection over the surgical site and liver while remaining 20 ml at the end of procedure after securing haemostasis over gall bladder bed and liver.
  Interventions: Drug: Ketamine
- Group B (Active Comparator): In Group B, bupivacaine 2mg/kgdiluted in normal saline to a total volume of 40ml .
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Ketamine — In Group K, ketamine 0.25mg/kg diluted in normal saline to a total volume of 40 ml was instilled by the surgeon, 20 ml before starting gall bladder dissection over the surgical site and liver while remaining 20 ml at the end of procedure after securing haemostasis over gall bladder bed and liver.
  Arms: Group K
Drug: Bupivacaine — In Group B, bupivacaine at a dose of 2 mg/kg was diluted in normal saline to a total volume of 40 ml. The administration was performed by the surgeon in two stages: the first 20 ml was instilled before starting the gall bladder dissection, applied over the surgical site and liver, while the remaining 20 ml was instilled at the end of the procedure after achieving hemostasis, applied over the gall bladder bed and liver.
  Other Names: Active compitator
  Arms: Group B

SUMMARY:
The intraperitoneal approach is used in anesthesia to manage the pain associated with abdominal procedures. Few studies have been conducted comparing intraperitonela ketamine with bupivacaine for pain control in laparoscopic cholecystectomy (LC) patients. To compare effect of intraperitoneal ketamine versus bupivacaine for postoperative pain control after LC. Department of Anesthesiology, Critical Care and Pain Management, Liaquat National Hospital and Medical College, Karachi. Group K received ketamine whereas Group B received bupivacaine. In Group K, ketamine 0.25mg/kg diluted in normal saline to a total volume of 40 ml was instilled by the surgeon. In Group B, bupivacaine 2mg/kgdiluted in normal saline to a total volume of 40ml was administered. Tramadol 1.5 mg/kg to a maximum of 100 mg IV was given as rescue analgesia. The pain was assessed using a numeric rating scale (NRS) with zero being no pain to ten being the worst possible pain. Pain was assessed using NRS at 0 hour (immediate postoperative period), 2 hour, 4 hour, 6 hour and 12 hours postoperatively.

DETAILED DESCRIPTION:
Proper pain management encourages quick ambling, reduces the likelihood of pulmonary embolism and deep vein thrombosis, enhances the patient's ability to breathe deeply, which reduces the possibility of pulmonary complications, and reduces tachycardia and the unnecessary investigations that are linked to it. Few studies have been conducted comparing intraperitoneal ketamine with bupivacaine for pain control in LC patients. Thus we planned the current study to compare effect of intraperitoneal ketamine versus bupivacaine for post-surgery pain control after LC.

This double blinded randomized controlled trial was performed in Operation theatre, Department of Anesthesiology, Critical Care and Pain Management, Liaquat National Hospital and Medical College, Karachi, Pakistan. The study was commenced with the institutional ethical approval. The study included all ASA I and II patients, male or female, aged 20 to 70, who were planned to undergo elective LC. Patients with known allergies to study drugs with any chronic pain condition, taking chronic pain medications, having psychiatric illness, weighing more than 80 kg, emergency surgery and converted to open cholecystectomy were excluded. Patients were enrolled with their written informed consent.

Sample size of 46 per arm was estimated using online available calculator Open-Epi, by taking mean VAS score of 3.0±0.86 in ketamine group and 3.50±0.84 in bupivacaine group at 12 hour at power of 80% and 95% confidence interval. Patients were enrolled using a consecutive sampling procedure, while groups were assigned at random using opaque, sealed envelopes that were consecutively numbered.

In Group K, ketamine 0.25mg/kg diluted in normal saline to a total volume of 40 ml was instilled by the surgeon, 20 ml before starting gall bladder dissection over the surgical site and liver while remaining 20 ml at the end of procedure after securing haemostasis over gall bladder bed and liver. In Group B, bupivacaine 2mg/kg diluted in normal saline to a total volume of 40ml was administered in similar way as described in Group K.

Patients' demographic profile including age, gender, body mass index (BMI), clinical profile comorbidity, ASA grade, surgery duration and pain status were documented. Weight (kg) divided by the square of height (m) was the definition of BMI. Co-morbidities of patients was confirmed from previous medical records or evidence against medication to treat underlying condition.

ELIGIBILITY:
Inclusion Criteria:

* Patients of age 20-70 years
* Patients of either gender
* Patients planned to undergo elective LC

Exclusion Criteria:

* Patients known to allergic to study drugs
* Patients with chronic pain conditions
* Patients taking chronic pain medications
* Patients having psychiatric illness
* Patients weighing more than 80 kg,
* Emergency surgery and/or converted to open cholecystectomy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
pain status | 2 hour, 4 hour, 6 hour and 12 hours postoperatively.
  The pain was assessed using a numeric rating scale (NRS) with zero being no pain to ten being the worst possible pain. Pain was assessed using NRS at 0 hour (immediate postoperative period), 2 hour, 4 hour, 6 hour and 12 hours postoperatively.

CONTACTS AND LOCATIONS:
Locations (1):
- Liaquat National Hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ziaei P, Kargar S, Dehghan MH, Madadizadeh F, Jamshidi HR. Clinical Trial of Intraperitoneal Administration of Ketamine Combined with Bupivacaine on Pain Status after Laparoscopic Cholecystectomy. Journal of Shahid Sadoughi University of Medical Sciences. 2022.
- [Background] Mostafa, R.H. and Mekki, Y.M.H., 2018. Comparative evaluation of intraperitoneal bupivacaine and bupivacaine ketamine combined with lung recruitment for reducing postoperative shoulder pain in laparoscopic cholecystectomy. Egyptian Journal of Anaesthesia, 34(4), pp.159-164.
- [Background] Moharari RS, Hadavi M, Pourfakhr P, Najafi A, Etezadi F, Khajavi MR. Evaluation of the postoperative analgesic efficacy of intraperitoneal ketamine compared with bupivacaine in laparoscopic cholecystectomy. Arch Anesthesiol Crit Care. 2016;2(1):146-9.